CLINICAL TRIAL: NCT05344313
Title: Oral Nutritional Supplementation With HMB Enhance Muscle Quality in Sarcopenic Surgical Patients (HEROS) - a Pilot Interventional Cohort Study
Brief Title: Oral Nutritional Supplementation With HMB Enhance Muscle Quality in Sarcopenic Surgical Patients
Acronym: HEROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Koh Hong Xiang Frederick, Principal Investigator, Consultant Colorectal Surgeon, Sengkang General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/2027
Record Dates: First submitted 2022-04-03; First posted 2022-04-25 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Frailty
Keywords: Nutrition; Prehabilitation; Surgery; Rehabilitation; Exercise; HMB
MeSH Terms: conditions — Sarcopenia; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: interventional cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sarcopenic patients (Experimental): Ensure Plus Advance + resistance training (Prehab) Rehabilitation 2months post surgery
  Interventions: Dietary Supplement: Ensure Plus Advance
- Healthy individuals (No Intervention): To make meaningful comparison of muscle quality, 10 healthy non-sarcopenic individuals from the same age range would also be recruited and will undergo muscle quality assessment using MuscleSound® once upon recruitment so that an objective comparison for IMAT can be made with our sarcopenic study cohort. This is to aid the study team to identify "normal" IMAT vs an IMAT for sarcopenic individuals. Any improvement of our cohort's muscle quality can be benchmarked against healthy muscle quality so that more meaningful comparison can be made. This control group would not be undergoing surgery, nor will they have any ONS supplied.

INTERVENTIONS:
Dietary Supplement: Ensure Plus Advance — as in the arm description of the intervention
  Other Names: Resistance training+2 months of rehabilitation
  Arms: Sarcopenic patients

SUMMARY:
Aims:

Clinical frailty severely impacts the physical, functional and physiological reserves necessary for the recovery after surgery. Sarcopenia, a multifactorial, multi-organ process which lead to loss of muscle mass over time, eventually resulting in clinical frailty. These 2 entities result in an increased morbidity and mortality from surgery. They also lead to a slower recovery from surgery with some patients never reaching baseline function after their surgery. It is, therefore, important to optimize patients with sarcopenia prior to surgery to reduce the incidence of morbidity and mortality.

Nutrition and resistance training have been shown to be able to curb the effects of sarcopenia. However, the type and regime of nutrition is still unknown.

Hypotheses:

The study team hypothesize that Ensure Plus Advance + HMB (beta-hydoxy-beta-methylbutyrate) would reduce the amount of IMAT (inter and intramuscular adipose tissue) in sarocpaenic patients after 2-4 weeks of prehabilitation. This effect would be sustained even after surgery and would continue to improve up to 3-months post-surgery whilst participating in rehabilitation. Taking Ensure Plus Advance + HMB would also improve functional parameters after prehabilitation, ensure a similar QoL 1-month post-surgery even if biochemical parameters may not show a significant improvement.

Methods:

The investigators would be conducting a pilot interventional cohort with an institution with an established prehabilitation programme (SKH) to evaluate the effect of the use a high protein, high calorie oral nutritional supplement (ONS) with HMB on muscle quality, using a device with Automated Intelligence (AI), in sarcopenic patients undergoing gastrointestinal surgery. Primary outcomes will be changes in Intermuscular Adipose Tissue (IMAT) while secondary outcomes include changes in functional parameters, quality-of-life (QoL), surgical outcomes and biochemical results.

ELIGIBILITY:
Inclusion Criteria:

1. between 40-90 years old
2. are sarcopenia (defined by the Asian Workgroup of Sarcopenia 2019 definition)
3. due to undergo elective major gastrointestinal surgery
4. able to satisfy at least 2 weeks of prehabilitation before surgery
5. ambulant
6. able to comply with physiotherapy and dietician advice

Exclusion Criteria:

1. Are pregnant
2. Are prisoners
3. Intellectually, mentally or emotionally deemed not able to provide an informed consent and/or are unable to fill up the post-procedure questionnaires
4. Have disease conditions requiring emergent/semi-emergent operation
5. Diabetes on oral hyperglycemic agents (OHGA)
6. Chronic Kidney Disease (CKD) or End-stage Renal Failure (ESRF)
7. Unable to or decline assessment for sarcopenia

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
change of Inter-muscular adipose tissue (%) between baseline and 1 day before surgery | 1 day before surgery
  change of Inter-muscular adipose tissue (%) between baseline and 1 day before surgery

SECONDARY OUTCOMES:
Change of handgrip strength after the prehabilitation programme | 1 day before surgery
  Change of handgrip strength after the prehabilitation programme
Change of gait speed after the prehabilitation programme | 1 day before surgery
  Change of gait speed after the prehabilitation programme
change in average length of hospitalization | up to 30 days post surgery
  change in average length of hospitalization
change of Inter-muscular adipose tissue (%) from pre-surgery to 3-months post-surgery | 3 months post surgery
  change of Inter-muscular adipose tissue (%) from pre-surgery to 3-months post-surgery
change in quality of life measure (EuroQol-5D) at 1-, 2- and 3-months post-surgery | 1,2 and 3 months post surgery
  change in quality of life measure (EuroQol-5D) at 1-, 2- and 3-months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frederick H Koh, FRCSEd, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Prevailing PDPA and HBRA regulations does not allow for open sharing. However, anonymised data can be shared if specifically requested for.